CLINICAL TRIAL: NCT04632134
Title: Long-term Effects of Transcutaneous Vagal Nerve Stimulation on Symptoms and Cardiovascular Autonomic Profile of Patients With Postural Orthostatic Tachycardia Syndrome (POTS)
Brief Title: Long-term Effects of Transcutaneous Vagal Nerve Stimulation on Postural Orthostatic Tachycardia Syndrome (POTS)
Acronym: VAG-POTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111
Record Dates: First submitted 2019-09-04; First posted 2020-11-17 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2021-06

CONDITIONS: Orthostatic Intolerance; Postural Tachycardia Syndrome; Syncope, Postural; Physical Disability; Autonomic Dysfunction
Keywords: Postural Orthostatic Tachycardia Syndrome; Vagal stimulation; Heart Rate
MeSH Terms: conditions — Orthostatic Intolerance; Postural Orthostatic Tachycardia Syndrome; Syncope; Primary Dysautonomias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous vagal nerve stimulation (tVNS) (Experimental): After positioning the tVNS electrodes in the right ear but without delivering tVNS (Sham tVNS), above mentioned signals will be recorded for 10 minutes while supine, for 15 minutes during 75° head-up tilt.
  The same protocol will be performed during active tVNS.
  The tVNS will be performed while 15 minutes in supine position and during 75°head-up Tilt.
  Thereafter, every patient will be provided with a Nemos© device and electrodes for home daily stimulation. Daily stimulation will consist of 4 hours of stimulation organized as 4 sessions each lasting 1 hour, to be applied at the patient's convenience.
  Interventions: Device: Transcutaneous vagal nerve stimulation (tVNS); Other: Placebo; Device: Home daily transcutaneous vagal nerve stimulation

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation (tVNS) — Transcutaneous vagal nerve stimulation (tVNS) will be performed using a noninvasive battery powered Transcutaneous Electrical Nerve Stimulation device (Nemos ©; Cerbomed, Germany). Electrical stimulation will be delivered by external electrodes through the skin surface at the conca of right external ear. Electrical current will be applied continuously with a pulse width of 200 μs and pulse frequency of 25 Hz. Stimulation amplitude will be adjusted between 0.1-6 mA, to a maximal amplitude level without causing patient discomfort.
  Other Names: Transcutaneous Electrical Nerve Stimulation device (Nemos ©; Cerbomed, Germany) European Conformity (CE) marking n°0408
Other: Placebo — tVNS electrodes will be positioned in the right ear of the POTS patients without delivering stimulus (Sham)
  Other Names: Sham stimulation
Device: Home daily transcutaneous vagal nerve stimulation — The home stimulation will consist of 4 hours of stimulation by the tVNS device organized as a 4 sessions of 1 hour. The home stimulation will last for 14 consecutive days.

SUMMARY:
Postural Orthostatic Tachycardia Syndrome (POTS) is characterized by symptoms of chronic orthostatic intolerance such as fatigue, lightheadedness, dizziness, palpitations and by pronounced tachycardia upon standing.

The aims of the present research study are to test whether a daily transcutaneous vagal nerve stimulation (tVNS) performed for 14 consecutive days may improve heart rate response and reduce disabling symptoms while standing.

DETAILED DESCRIPTION:
Postural Orthostatic Tachycardia Syndrome (POTS) is characterized by symptoms of chronic orthostatic intolerance such as fatigue, lightheadedness, dizziness, palpitations and by pronounced tachycardia without hypotension upon standing. In healthy volunteers, transcutaneous vagal nerve stimulation (tVNS) may result in increased cardiac vagal activity and reduced vascular sympathetic drive with minimal, if any, side effects. It is possible to hypothesize that any therapeutic intervention aimed at increasing cardiac vagal modulation might result in clinical improvement of the disease.

The aim of the study are to evaluate the medium-term effects of tVNS, performed every day for a 14 days on cardiovascular autonomic profile and symptoms intensity in POTS patients.

Study and General Design

Phase 1- Enrollment:

23 POTS patients, older than 18 years of age, will be consecutively enrolled. Each POTS patient will undergo complete medical evaluation at the time of enrollment, which will take place seven days before baseline recordings (i.e. Control day, see below), in order to individually optimize the tVNS amplitude and get patients familiarized with both the tVNS procedure and the clinical laboratory environment. On the same day, 30-minute continuous tVNS will be delivered to the patients under rigorous medical and hemodynamic supervision to exclude any kind of short term adverse effects.

Transcutaneous vagal nerve stimulation (tVNS) will be performed using a noninvasive battery powered Transcutaneous Electrical Nerve Stimulation device (Nemos ©; Cerbomed, Germany). Electrical stimulation will be delivered by external electrodes through the skin surface at the conca of right external ear. Electrical current will be applied continuously with a pulse width of 200 μs and pulse frequency of 25 Hz, differently from previous protocols. Stimulation amplitude will be adjusted between 0.1-6 milliampere (mA), to a maximal amplitude level without causing patient discomfort.

Phase 2 Sham tVNS and Effective tVNS:

In every subject continuous ECG, beat by beat non-invasive arterial pressure (Nexfin device), respiratory activity by thoracic piezoelectric belt will be recorded while supine and during 75° head-up tilt (rest-tilt protocol). After positioning the tVNS electrodes in the right ear but without delivering tVNS (Sham tVNS), above mentioned signals will be recorded for 10 minutes while supine, for 15 minutes during 75° head-up tilt. The same protocol will be repeated during stimulation amplitude will be adjusted to maximal tolerable level as assessed in Phase 1 (effective acute tVNS).

The Composite Autonomic Symptom Scale (COMPASS 31) COMPASS 31 will be used to quantify the following autonomic symptoms: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, urinary and pupillomotor dysfunction symptoms .

Phase 3-Home daily stimulation:

Thereafter, every patient will be provided with a Nemos© device and electrodes for home daily stimulation. Daily stimulation will consist of 4 hours of stimulation organized as 4 sessions each lasting 1 hour, to be applied at the patient's convenience.

Phase 4- Post- 14-day tVNS. After 14 days of home daily tVNS, all the patients will undergo the rest-tilt protocol described in Phase 2.

COMPASS 31 questionnaire will be administered while supine and during 75° head-up Tilt

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Postural Orthostatic Tachycardia Syndrome
* Older than 18 years

Exclusion Criteria:

* Dysautonomias other than POTS
* Neurodegenerative diseases
* History/family history of seizures
* Atrial fibrillation and other relevant cardiac rhythm disturbances
* Chronic inflammatory diseases
* Chronic use on anti-inflammatory drugs
* Diabetes
* Other neurological or psychiatric diseases
* Pacemakers or other electronic implants inserted into the body
* Coronary disorders
* Elevated intracranial blood pressure
* Assumption of drugs facilitating seizures
* Assumption ofpsychiatric drugs
* Alcohol abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Estimated)
Dates: Start 2019-11-10 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Autonomic symptoms | Change from baseline Autonomic symptoms at 14 days
  Autonomic symptoms will be assessed by the Composite Autonomic Symptom Scale (COMPASS 31) questionnaire. This is based on 31 items and a score ranging from 0 to100, 0 being the absence of symptom and 100 the greatest symptom intensity. The COMPASS 31 will be used to quantify the following autonomic symptoms: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, urinary and pupillomotor dysfunction symptoms.

SECONDARY OUTCOMES:
Change in Heart rate | Change from baseline cardiovascular autonomic profile at 14 days
  Change of Cardiovascular autonomic profile
Change in blood pressure | Change from baseline cardiovascular autonomic profile at 14 days
  Change of Cardiovascular autonomic profile
Change in respiration rate | Change from baseline cardiovascular autonomic profile at 14 days
  Change of Cardiovascular autonomic profile

CONTACTS AND LOCATIONS:
Overall Officials: Raffaello Furlan, Prof, Study Director — Humanitas Research Hospital; Humanitas University; Franca Barbic, MD, Study Chair — Humanitas Research Hospital; Humanitas University; Dana Shiffer, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Humanitas Research Hospital, Rozzano, Italy

REFERENCES:
- [Background] Raj SR. Postural tachycardia syndrome (POTS). Circulation. 2013 Jun 11;127(23):2336-42. doi: 10.1161/CIRCULATIONAHA.112.144501. No abstract available. PMID 23753844
- [Background] Robertson D. The epidemic of orthostatic tachycardia and orthostatic intolerance. Am J Med Sci. 1999 Feb;317(2):75-7. doi: 10.1097/00000441-199902000-00001. No abstract available. PMID 10037110
- [Background] Furlan R, Jacob G, Snell M, Robertson D, Porta A, Harris P, Mosqueda-Garcia R. Chronic orthostatic intolerance: a disorder with discordant cardiac and vascular sympathetic control. Circulation. 1998 Nov 17;98(20):2154-9. doi: 10.1161/01.cir.98.20.2154. PMID 9815870
- [Background] Clancy JA, Mary DA, Witte KK, Greenwood JP, Deuchars SA, Deuchars J. Non-invasive vagus nerve stimulation in healthy humans reduces sympathetic nerve activity. Brain Stimul. 2014 Nov-Dec;7(6):871-7. doi: 10.1016/j.brs.2014.07.031. Epub 2014 Jul 16. PMID 25164906
- [Background] Napadow V, Edwards RR, Cahalan CM, Mensing G, Greenbaum S, Valovska A, Li A, Kim J, Maeda Y, Park K, Wasan AD. Evoked pain analgesia in chronic pelvic pain patients using respiratory-gated auricular vagal afferent nerve stimulation. Pain Med. 2012 Jun;13(6):777-89. doi: 10.1111/j.1526-4637.2012.01385.x. Epub 2012 May 8. PMID 22568773
- [Background] Fu Q, Vangundy TB, Galbreath MM, Shibata S, Jain M, Hastings JL, Bhella PS, Levine BD. Cardiac origins of the postural orthostatic tachycardia syndrome. J Am Coll Cardiol. 2010 Jun 22;55(25):2858-68. doi: 10.1016/j.jacc.2010.02.043. PMID 20579544
- [Background] Murray AR, Atkinson L, Mahadi MK, Deuchars SA, Deuchars J. The strange case of the ear and the heart: The auricular vagus nerve and its influence on cardiac control. Auton Neurosci. 2016 Aug;199:48-53. doi: 10.1016/j.autneu.2016.06.004. Epub 2016 Jun 28. PMID 27388046
- [Background] Furlan R, Porta A, Costa F, Tank J, Baker L, Schiavi R, Robertson D, Malliani A, Mosqueda-Garcia R. Oscillatory patterns in sympathetic neural discharge and cardiovascular variables during orthostatic stimulus. Circulation. 2000 Feb 29;101(8):886-92. doi: 10.1161/01.cir.101.8.886. PMID 10694528
- [Background] Low PA. Composite autonomic scoring scale for laboratory quantification of generalized autonomic failure. Mayo Clin Proc. 1993 Aug;68(8):748-52. doi: 10.1016/s0025-6196(12)60631-4. PMID 8392653